CLINICAL TRIAL: NCT00299754
Title: The Randomised-Controlled Trial Of Misoprostol And Dinoprostone Vaginal Pessaries for Cervical Priming (TROMAD Study)
Brief Title: Trial Of Misoprostol And Dinoprostone Vaginal Pessaries for Cervical Priming (TROMAD Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National Healthcare Group, Singapore (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TCTan001
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2006-03-07 (Estimated); Status verified 2005-06

CONDITIONS: Induction of Labour
Keywords: Low dose misoprostol; dinoprostone; cervical priming
MeSH Terms: interventions — Misoprostol

INTERVENTIONS:
Drug: Misoprostol

SUMMARY:
Most studies of labour induction with misoprostol used doses higher than 25mg and intervals of 3-4 hours. We studied a low-dose regime of 25mg misoprostol and compared its efficacy as single dose or double dose with dosing interval of 6 hours to our current regime of 3 mg dinoprostone pessary.

DETAILED DESCRIPTION:
171 women with singleton term pregnancies and modified Bishop score (mBS) ≤ 5 were recruited and randomized into 3 arms: current dinoprostone regime, double dose misoprostol or single dose misoprostol. The primary outcome was the number of women who achieved favourable mBS>6 or active labour by Day 2. Secondary outcomes were time interval from insert to active labour or delivery, abnormal uterine activity, delivery method and adverse neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy, cephalic presentation, gestation greater than 37 completed weeks, no known contraindication to vaginal delivery, and Bishop score≤5.

Exclusion Criteria:

* previous caesarean section or other uterine surgery, significant maternal medical/obstetric complication in pregnancy (such as severe pre-eclampsia, significant antepartum haemorrhage), antepartum evidence of fetal compromise (such as fetal growth restriction), previous attempt at cervical priming, contraindication to receiving prostaglandins, including asthma and glaucoma.

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 171
Dates: Start 2003-01; Study Completion 2004-12

PRIMARY OUTCOMES:
The primary outcome was the number of women who achieved favourable mBS>6 or active labour by Day 2.

SECONDARY OUTCOMES:
Secondary outcomes were time interval from insert to active labour or delivery, abnormal uterine activity, delivery method and adverse neonatal outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Thiam-Chye Tan, Principal Investigator — KK Women's and Children's Hospital; Tseng-Meng Chua, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Result] Rath W. A clinical evaluation of controlled-release dinoprostone for cervical ripening--a review of current evidence in hospital and outpatient settings. J Perinat Med. 2005;33(6):491-9. doi: 10.1515/JPM.2005.087. PMID 16318611